CLINICAL TRIAL: NCT00000396
Title: Evaluating/Reinforcing Arthritis Patient Education for Urban African Americans
Brief Title: Arthritis Patient Education for Urban African Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Larry Gruppen, Professor of Medical Education, University of Michigan
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: P60AR020557 (NIH); P60AR020557 (NIH); NIAMS-016
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Arthritis
Keywords: Arthritis; Arthritis education; African Americans; Self-help; Self-management; Cultural beliefs
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Education in Arthritis Self-Help Course
  Interventions: Behavioral: Patient self-care education

INTERVENTIONS:
Behavioral: Patient self-care education

SUMMARY:
Research has shown that people with arthritis can improve their ability to cope with arthritis pain with the help of patient education programs, which teach people things they can do to help manage their disease. However, we do not know much about the effects of arthritis patient education programs on minorities, such as urban African Americans.

We will gather participants for this project through a faith-based community network. The project is made up of four studies that will provide information about culturally relevant ways of reaching urban African Americans with arthritis and providing patient education that addresses arthritis care needs of the African American community. This project will also provide information on the effectiveness of an arthritis self-help course for urban African Americans. We hope to better understand the differences among cultural groups and how these differences should affect the design of culturally appropriate patient education.

DETAILED DESCRIPTION:
Clinical studies have shown that arthritis patient education interventions are an effective addition to medical treatment in improving patients' ability to cope with pain, thereby reducing perceived symptom severity, improving patients' ability to help themselves, and providing them with skills and strategies for dealing with limits on daily activities. We know little, however, about generalizing the effects of such programs to cultural minority groups, such as urban African Americans. We know even less about the longevity of any benefits of patient education or about effective reinforcement and maintenance techniques. To examine these issues, we will recruit participants for this project through a faith-based community network to pursue the following aims:

1. Evaluate the impact of arthritis patient education on arthritis symptoms and pain levels, functional status, self-care knowledge and behaviors, self-efficacy, emotional status, and health care resource use through a randomized controlled trial (Study 1).
2. Test the impact of focused reinforcement of the concepts in the Arthritis Self-Help Course (ASHC) over a 12-month period through a randomized controlled trial (Study 2).
3. Examine the detailed educational dynamics of the ASHC, identify aspects of the course that are less effective with or relevant to African Americans, and identify modes of communication and presentation used in the course that require adaptation for an African American audience (Study 3).
4. Assess the personal and cultural belief systems underlying African Americans' understanding of arthritis and their use of conventional and unconventional arthritis treatments (Study 4).

These studies will provide valuable information regarding culturally relevant methods of reaching urban African Americans with arthritis and providing patient education that addresses arthritis care needs of the African American community. This study will also clarify the longevity of educational benefits and the effectiveness of alternative methods of educational reinforcement in this population. The exploratory studies of individual beliefs and knowledge of arthritis and its treatment, and the formal evaluation of a patient education program, will provide a better understanding of the ways in which cultural groups differ and how these differences should influence the design and delivery of culturally appropriate patient education.

ELIGIBILITY:
Inclusion Criteria:

* Urban African Americans with arthritis
* 18 years or older

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 1997-09; Primary Completion 2001-03 (Actual); Study Completion 2002-10 (Actual)

PRIMARY OUTCOMES:
Knowledge of arthritis self-care behaviors | Measured upon completion of the educational intervention and at 6-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Larry D. Gruppen, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States